CLINICAL TRIAL: NCT03333031
Title: A Phase I Study of HS-196, an HSP90 Inhibitor-linked Near Infrared Probe for Detection of Solid Malignancies
Brief Title: A Study of HS-196, an HSP90 Inhibitor-linked NIR Probe for Solid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding ended
Sponsor: Herbert Lyerly (Other)
Responsible Party: Sponsor-Investigator, Herbert Lyerly, Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00082272
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Solid Tumor
Keywords: cancer; imaging agent; HSP90
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HS-196 (Experimental): HS-196 will be administered intravenously as a single dose
  Interventions: Drug: HS-196

INTERVENTIONS:
Drug: HS-196 — HS-196 will be administered intravenously as a single dose

SUMMARY:
HS-196 is near infrared red (NIR)-tethered HSP90 inhibitor for clinical imaging of selective tumor binding. HS-196 consists of a HSP90 inhibitor that binds competitively to the Hsp90 ATP binding domain connected by a linker to a contrast agent (near infrared (NIR) dye) that can be used for imaging. HS-196 can freely enter tumor cells to selectively bind Hsp90. Due to the the NIR dye, HS-196 accumulation in the malignant cells allows for specific visualization of tumors within the body.

DETAILED DESCRIPTION:
The product to be tested under this IND, HS-196, is a tumor imaging agent.

Hsp90 (heat shock protein 90) is a chaperone protein that aids in the folding, stabilization, and degradation of cellular proteins and is found in virtually all living organisms. Cancer cells in particular have high expression of Hsp90. Hsp90 has three structural domains including an N-terminal domain that contains an ATP binding site. Small molecule inhibitors of HSP90 (Hsp90i) can selectively and competitively to the Hsp90 ATP binding domain. HS-196 consists of a HSP90 inhibitor that binds competitively to the Hsp90 ATP binding domain connected by a linker to a contrast agent (near infrared (NIR) dye) that can be used for imaging. HS-196 can freely enter tumor cells to selectively bind Hsp90. Due to the the NIR dye, HS-196 accumulation in the malignant cells allows for specific visualization of tumors within the body.

HS-196 will be used in this investigation for the imaging of solid tumors The objectives of the study are to determine the dose of HS-196 that achieves the greatest ratio of tumor to normal tissue fluorescence in patients with malignancy, the safety of HS-196 administration in patients with malignancy, the average radiant efficiency in resected tumors following HS-196 administration, the localization of the HS-196 by microscopy of tumor slices, and the PK metrics of HS-196 when administered to patients.

ELIGIBILITY:
Inclusion Criteria:

For Dose escalation and recommended dose phases:

* Diagnosis of a solid malignancy, stage I-IV, with planned surgical resection or biopsy.

For Expansion phase:

* Patients with mammographically detected breast nodules with planned surgical resection or biopsy.

For All phases:

* ECOG 0 or 1
* Estimated life expectancy > 3 months
* Age ≥ 18 years
* Adequate hematologic function, with WBC ≥ 3000/microliter, hemoglobin ≥ 9 g/dL (it is acceptable to have had prior transfusion), platelets ≥ 75,000/microliter; PT-INR <1.5, PTT <1.5X ULN
* Adequate renal and hepatic function, with serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL), ALT and AST ≤ 2.5 x upper limit of normal or if liver metastases are present < 5 x upper limit of normal.
* Female patients must be of non-child-bearing potential or use effective contraception, e.g., use of oral contraceptives with an additional barrier method (since the study drug may impair the effectiveness of oral contraceptives), double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), Depo-Provera, partner vasectomy, total abstinence, and willing to continue the effective contraception method for 30 days after the last dose of study drug;
* Ability to understand and provide signed informed consent that fulfills Institutional Review Board's guidelines.
* Ability to return to Duke University Medical Center for adequate follow-up, as required by this protocol.

Exclusion Criteria:

* Serious chronic or acute illness considered by the P.I. to constitute an unwarranted high risk for investigational drug treatment.
* Medical or psychological impediment to probable compliance with the protocol.
* Asthma under medical management
* Uncontrolled high blood pressure
* Presence of a known active acute or chronic infection including HIV or viral hepatitis (Hepatitis B and C)).
* Pregnant or nursing women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Fluorescence | 1 day
  Ratio of tumor to normal tissue fluorescence

SECONDARY OUTCOMES:
Number of AEs | 1 month
  Safety of HS-196 administration in patients with malignancy
Radiant Efficiency | 1 day
  The average radiant efficiency in resected tumors following HS-196 administration.
HS-196 Localization | 1 day
  Localization of the HS-196 by microscopy of tumor slices.
Maximum Plasma concentration Cmax | 1 week
  PK metrics of HS-196 when administered IV to patients
Area Under the Curve AUC | 1 week
  PK metrics of HS-196 when administered IV to patients

CONTACTS AND LOCATIONS:
Overall Officials: H. Kim Lyerly, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided